CLINICAL TRIAL: NCT01170429
Title: A Multicentered, Double-blinded, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Procaterol Hydrochloride With Inhaled Glucocorticoid in Treatment Patients With Cough Variant Asthma (CVA)
Brief Title: Efficacy and Safety Study of Procaterol Hydrochloride to Treat Patients With Cough Variant Asthma (CVA)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Xin Zhou/Director of Respiratory Department, Shanghai Jiao Tong University Affiliated 1st People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002-ZOC-0902i
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-06

CONDITIONS: Cough Variant Asthma
Keywords: Cough Variant Asthma; Procaterol Hydrochloride
MeSH Terms: conditions — Cough-Variant Asthma | interventions — Procaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I. Procaterol Hydrochloride (Experimental): Meptin (Procaterol hydrochloride) Tablets, 25µg twice daily orally plus inhaled budesonide 200µg twice daily for eight weeks;
  Interventions: Drug: Procaterol hydrochloride
- II. Procaterol hydrochloride placebo (Placebo Comparator): Meptin placebo (Procaterol hydrochloride) Tablets, 25µg twice daily orally plus inhaled budesonide 200µg twice daily for eight weeks;
  Interventions: Drug: Meptin placebo

INTERVENTIONS:
Drug: Procaterol hydrochloride — 25µg BID for 8 weeks
  Other Names: Meptin
  Arms: I. Procaterol Hydrochloride
Drug: Meptin placebo — 25µg BID for 8 weeks
  Other Names: Meptin
  Arms: II. Procaterol hydrochloride placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of procaterol hydrochloride with inhaled glucocorticoid in treatment patients with cough variant asthma (CVA).

DETAILED DESCRIPTION:
This is a 8-week, double-blind, randomized, placebo-controlled study, the patients with CVA will be randomized to experimental or placebo control group.

During the screening period, eligible patients will be evaluated by cough symptom score and LCQ life quality score. After 4 and 8 weeks treatment, patients will be evaluated by cough symptom score and LCQ life quality score respectively. Adverse events will also be captured at every visit.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients,18-75 years old;
* cough lasting over 3 weeks ; dry cough or with slight white mucous phlegm; cough is the main clinical symptom or the only symptom;
* without wheeze and fever;
* without the history of upper respiratory tract infection within recent two months; non-smoking or giving-up smoking for over two years;
* without rales from lung;
* no obvious abnormalities from chest X-ray;
* bronchial provocation test: positive.

Exclusion Criteria:

* patients with chronic pulmonary disease;
* patients who are allergic to ß2 receptor agonist;
* patients taking ß2 receptor agonist for long time;
* severe heart, renal and hepatic disease;
* unable to comply with the protocol;
* pregnant, breast feeding, and childbearing potential women;
* patients improper to the trial according to the investigators' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Patient cough symptom score | 8 weeks
Therapy duration | 8 weeks
Rates of adverse events | 8 weeks

SECONDARY OUTCOMES:
LCQ Life Quality Score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zhou, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xin Zhou, Shanghai, Shanghai Municipality, China